CLINICAL TRIAL: NCT03618485
Title: Registry of Patients With Myeloproliferative Neoplasms (MPNs) in Taiwan -Taiwan MPN Working Group
Brief Title: Registry of Patients With MPNs in Taiwan
Status: Active, not recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Lee-Yung Shih, Clinical Professor, Chang Gung Memorial Hospital
Other Study IDs: 201700356B0
Record Dates: First submitted 2018-07-16; First posted 2018-08-07 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Myeloproliferative Neoplasms
MeSH Terms: conditions — Myeloproliferative Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Myeloproliferative neoplasms (MPNs) are a group of clonal hematologic malignancies with great variation in reported patient life expectancy and are characterized by a relatively indolent course which can be complicated by thromboembolic events and transformation to acute myeloid leukemia (AML).

The MPNs in the 2016 World Health Organization (WHO) classification of myeloid neoplasms consist of polycythemia vera (PV), essential thrombocythemia (ET), primary myelofibrosis (PMF) including prefibrotic/early stage and over fibrotic stage, chronic myeloid leukemia, other (rare) disorders such as chronic neutrophilic leukemia and chronic eosinophilic leukemia and MPN unclassifiable (MPN-U).

The prevalence and genetic characteristics of patients with MPNs in Taiwan are still unknown. Molecular tests which are required for the diagnosis of MPNs are not available in many hospitals which hamper the accurate diagnosis and subtype classification of MPNs. Moreover, the information of current therapeutic strategy for MPNs in most medical centers in Taiwan is also not available. The purpose of this MPN registry is to collect clinical data, molecular characteristics, treatment details and response to therapy, occurrence of complications during the course, disease progression to secondary myelofibrosis from PV or ET and secondary AML (sAML) transformation as well as survival. The clinical and molecular data including the high molecular risk (HMR) genes will be examined and correlated with treatment outcomes in Taiwanese MPN patients.

The Molecular Diagnostic Laboratory at Chang Gung Memorial Hospital-Linkou is a College of American Pathologists (CAP)-accredited lab which provides high quality of molecular genetic tests for hematologic malignancies. The three driver gene mutations are the major criteria for the diagnosis of MPN, the methodologies of mutational analyses have been well set up for the clinical use in this lab. In addition, this lab is also equipped with facilities for the detection of mutated genes which were recently identified as HRM category (presence of any of ASXL1, EZH2, SRSF2, IDH1 or IDH2), and mutations of other epigenetic regulators or splicing factors.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged ≥ 20 years.
2. Patient who had a confirmed diagnosis according to the 2016 revised WHO criteria with a Ph (-) MPN.

Exclusion Criteria:

1. Patients do not fulfill the diagnostic criteria of MPN by WHO 2016 classification.
2. Patients unwilling to sign informed consent.

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with MPNs newly diagnosed and followed in Chang Gung Memorial Hospital and cooperative hospitals.Registry will be limited to patients newly diagnosed between 2016 and 2019. Newly diagnosed means having the first bone marrow biopsy within 12 months from diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Epidemiological data of MPNs in Taiwan | 24 month
  The prevalence of MPNs during the whole study period in Taiwan

SECONDARY OUTCOMES:
The frequencies of mutations of driver genes in Taiwanese patients with MPNs. | 24 months
  The frequencies of JAK2V617F or JAK exon12, CALR and MPL in each subtype of patient's with MPN during the two years of study period.
Treatment required | 36 months
  Date of phlebotomy and date of initiation of drug therapy
Change of symptoms from baseline using MPN-10 symptom assessment. | 36 months
  Change of symptoms from baseline in MPN-10 at different time points (V2-5) during the study period.
Occurrence of vascular events | 36 months
  Date of occurrence of thrombosis or bleeding during the study period.
Occurrence of secondary acute myeloid leukemia (sAML) | 36 months
  Date of the development of sAML
Overall survival | 36 months
  Time from diagnosis of MPN to last follow-up or date of death measured by months

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital-Linkou, Taoyuan District, State, Taiwan